CLINICAL TRIAL: NCT04881695
Title: Evaluation of Child Desire in Young Women With Premature Ovarian Failure
Acronym: DESIOP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210157; 2020-A02741-38 (Other: IDRCB)
Record Dates: First submitted 2021-04-29; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Premature Ovarian Failure (POF)
Keywords: Desire children, infertility, medical assisted procreation
MeSH Terms: conditions — Primary Ovarian Insufficiency; Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Women aged 18-26 years with congenital (Turner syndrome or other determined or undetermined genetic cause) or acquired (post-therapeutic)
  Interventions: Other: Questionary patients
- Controls: Women aged 18-26 years who do not have a condition that compromises their fertility
  Interventions: Other: Questionary controls

INTERVENTIONS:
Other: Questionary patients — The patients will answer 1 questionnaire consisting of 5 parts :
  * General (demographic information)
  * Desire for a child
  * Hospital Anxiety and Depression scale
  * Sexual life
  * Additional questions regarding medical care
  Groups: Patients
Other: Questionary controls — Witnesses will complete 1 survey containing 4 parts:
  * General (demographic information)
  * Desire to have a child
  * Hospital Anxiety and Depression scale
  * Sexual life
  Groups: Controls

SUMMARY:
Premature ovarian failure (POF) is a rare condition, affecting 1 in 10,000 women before age 20 and 1 in 1,000 women before age 30. The two main causes of POF are congenital and acquired.

Patients with POF who carry out the desire to have a child turn to medically assisted reproduction through oocyte donation or to adoption.

The main endpoint of this study is to compare the desire to have children among women with premature ovarian failure (POF) aged 18 to 26 years vs. controls of the same age (stratified by age) without major menstruation disorder.

DETAILED DESCRIPTION:
Premature ovarian failure (POF) is a rare condition, affecting 1 in 10,000 women before age 20 and 1 in 1,000 women before age 30. The two main causes of POF are congenital and acquired.

Patients with POF who carry out the desire to have a child turn to medically assisted reproduction through oocyte donation or to adoption.

The main endpoint of this study is to compare the desire to have children among women with premature ovarian failure (POF) aged 18 to 26 years vs. controls of the same age (stratified by age) without major menstruation disorder. The primary endpoint is the percentage of women with POF reporting a desire to have a child (yes / no) vs. controls of the same age with normal gonadal function/ The answers will be collected on two online questionnaires.

The secondary endpoints are:

* Look for a difference in the desire for a child according to the age at the diagnosis of POF, the cause of POF, the intake of hormone replacement therapy and the age of the patients at the time of the study.
* Assess the sexual life of women in POF.
* Assess the psychological state of women with POF-related infertility and help identify those with symptoms of anxiety or depression. He will be assessed by the Hospital Anxiety and Depression Questionnaire to help identify those with symptoms of anxiety or depression.

The women will be contacted by email and will receive a newsletter. The controls will be recruited from patients who have visited at least once at bicetre Hospital and who do not have a condition that could impair fertility. They must not have been pregnant or must not be pregnant at the time of the study. The email will contain a questionnaire.

We estimate that 120 patients will meet the inclusion and non-inclusion criteria among the patients on the Unit.

Considering that 80 patients (2/3) will answer the questionnaires, we will be able to include 80 patients and 80 controls in our study.

The proportion of women wishing to have children, in the general population, in the study age group is estimated at 90%. Including 160 participants will allow us to show a 20% difference in the proportion of desire to have children in patients with POF, with a power of 90%, an alpha risk of 5% and a bilateral formulation.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 26
* Diagnosed with POF according to the following criteria:

Absence of pubertal development or primary or secondary amenorrhea for more than 4 months Follicle Stimulating Hormone (FSH) rate> 40 mL U /L, on at least two separate samples taken at least one month apart Low estradiol level <40 pg / mL

* POF of congenital (Turner syndrome or other genetic cause) or acquired (post-therapeutic) origin
* Who consulted in the Adolescent and Young Adult Gynecology Unit at bicetre Hospital between 2014 and 2021

Exclusion Criteria:

* Minor patient or over 26 years old
* Inability to complete the questionnaire
* Lack of social security coverage
* Patient under state medical aid
* Patient under guardianship or curators or under legal protection
* POF not confirmed (for patients only)
* Condition impacting fertility or having already been pregnant or pregnant at the time of the study (for controls)

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Study Population: Women aged 18 to 26 with congenital POF (linked to Turner Syndrome or to another determined or undetermined genetic cause) or acquired (post-treatment), having consulted at least once at the bicetre hospital.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2021-05-10 (Estimated); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of POI patients expressing a desire for a child (yes/no) compared to controls of the same age with no fertility compromising condition, | 3 months
  To compare the desire for children of patients with premature ovarian failure (POI) aged 18-26 years with controls of the same age group (inclusion stratified by age in 2-year strata) with no fertility compromising condition.

SECONDARY OUTCOMES:
Assess the sexual life of women with POF | 3 months
  Assess the sexual life of women in POF by answering a questionary compared to the answers of controls.
  - The score of patients will be compared to the score of controls.
Assess the psychological state of women with POF-related infertility and help identify those with symptoms of anxiety or depression. | 3 months
  Assess by the Hospital Anxiety and Depression questionnaire to help identify those with symptoms of anxiety or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Lise DURANTEAU, Doctor, Principal Investigator — Hospital Bicetre
Locations (1):
- Hospital Bicetre, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No